CLINICAL TRIAL: NCT06124378
Title: Neoadjuvant Tislelizumab With Oxaliplatin and Capecitabine in Microsatellite Stable, Locally Advanced Colon Cancer (NETSAC): A Single-arm, Single-center, Exploratory Phase II Clinical Study
Brief Title: Neoadjuvant Tislelizumab With Chemotherapy for the Treatment of MSS Colon Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Minglin Lin
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Colonic Neoplasms; Neoadjuvant Therapy; Immune Checkpoint Inhibitors
Keywords: Colon cancer, Neoadjuvant chemotherapy; PD-1 inhibitor
MeSH Terms: conditions — Colonic Neoplasms | interventions — tislelizumab; Oxaliplatin; Capecitabine; Colectomy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab combined with Oxaliplatin and Capecitabine cohort (Experimental): Patients with locally advanced colon cancer who met the inclusion criteria received two or four cycles of Tislelizumab combined Capecitabine and Oxaliplatin regimen chemotherapy and were evaluated by enhanced CT. Then, these patients will receive curative surgery for colon cancer.
  Interventions:
  Drug: Oxaliplatin,130mg/m2 for chemotherapy on Day 1 every 3 weeks and repeat for 2 or 4 cycles.
  Drug: Capecitabine, Oral Capecitabine 1000 mg/m2 twice daily from Day 1 to Day 14 every 3 weeks and repeat for 2 or 4 cycles.
  Drug: Tislelizumab, 200 mg on Day 1 every 3 weeks and repeat for 2 or 4 cycles. Procedure: Colectomy
  Interventions: Drug: Tislelizumab; Drug: Oxaliplatin; Drug: Capecitabine; Procedure: Colectomy

INTERVENTIONS:
Drug: Tislelizumab — 200 mg on Day 1 every 3 weeks and repeat for 2 or 4 cycles. The incidence of adverse events with Tislelizumab is relatively low. The Tislelizumab dose adjustment was implemented according to the prescribing information.
  Other Names: Tevimbra
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 on Day 1 every 3 weeks and repeat for 2 or 4 cycles. The dose reduction protocol for oxaliplatin-induced toxicity was implemented according to the study in British Journal of Cancer (2018) 118:1322-1328.
  Other Names: Eloxatin
Drug: Capecitabine — Oral Capecitabine 1000 mg/m2 twice daily combined with oxaliplatin chemotherapy from Day 1 to Day 14 every 3 weeks and repeat for 2 or 4 cycles. The dose reduction protocol for capecitabine-induced toxicity was implemented according to the study in British Journal of Cancer (2018) 118:1322-1328.
  Other Names: Xeloda
Procedure: Colectomy — The specific surgical approach is laparoscopic. The tumor blood supply is ligated and cut at the root of the mesentery, and the margin of resection should be no less than 10cm. Complete resection of the mesocolon (CME) is performed in conjunction.
  Other Names: Surgery

SUMMARY:
This study aims to elucidate the effects of neoadjuvant Tislelizumab combined with chemotherapy in locally advanced Microsatellite Stable (MSS) colon cancer.

DETAILED DESCRIPTION:
The standard treatment for locally advanced colon cancer is complete mesocolic excision (CME) followed by adjuvant chemotherapy. The MOSAIC and 16968 studies have shown that about 30% of patients experience recurrence and metastasis within 6-7 years after surgery. Neoadjuvant chemotherapy may improve the prognosis of colon cancer patients. The significant tumor remission after neoadjuvant therapy probably indicates a better long-term survival for patients. The OPTICAL and Fluoropyrimidine Oxaliplatin and Targeted Receptor Pre-Operative Therapy (FoxTROT) studies have shown that approximately 35% of patients are resistant to oxaliplatin-containing neoadjuvant chemotherapy, with a pathological complete response (pCR) rate of less than 10% and uncertain survival improvement. Moreover, previous study shown that immunotherapy has unsatisfied efficacy for microsatellite stable (MSS) colon cancer. Therefore, it is necessary to explore more effective neoadjuvant treatment strategy for tumor therapy.

Immunogenic cell death will be enhanced by oxaliplatin-induced immunogenicity and combined with anti-programmed cell death 1 (PD-1) monoclonal antibodies for neoadjuvant therapy. The study will conduct 2 or 4 cycles of Tislelizumab with Oxaliplatin and Capecitabine, followed by CME surgery. The study's primary endpoint is the proportion of pCR in the pathological specimens of surgically resected tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤75 years old.
* Pathologically diagnosed MSS ((confirmed by microsatellite stable detection or next-generation target sequencing) or (confirmed by immunohistochemistry)) colon adenocarcinoma.
* The lower edge of the tumor is more than 12cm from the anus as measured by colonoscopy and the lower edge of the tumor cannot be directly palpated during rectal examination.
* Enhanced CT stage T4 or T1-4 N+ without multiple primary tumors or distant metastasis.
* The Eastern Cooperative Oncology Group physical status score is 0-1.
* Life expectancy is expected to be more than 1 year.
* First diagnosis, no previous anti-tumor treatment received, and no chemotherapy contraindications.
* Appropriate organ function is defined as follows: Hemoglobin level ≥ 60g/L, Neutrophil count ≥ 1.5×10^9/L, Platelet count ≥ 75×10^9/L, Serum total bilirubin ≤ 1.5× the upper limit of normal (UNL), Aspartate aminotransferase (AST) ≤ 2× UNL, Alanine aminotransferase (ALT) ≤ 3× UNL, Serum creatinine ≤ 1.5× UNL.
* Informed consent, able to understand the study protocol and willing to participate in the study, and will provide written informed consent.

Exclusion Criteria:

* Enhanced CT stage (T1-3N0M0)
* Multifocal colorectal cancer.
* CT or MRI in the mid-sagittal plane shows that the lower border of the tumor is below the line connecting the sacrococcygeal promontory and the upper border of the pubic symphysis.
* Tumor obstruction or high risk of obstruction, bleeding, and/or perforation requiring emergency surgery or stent placement.
* Cannot tolerate chemotherapy or immunotherapy, such as but not limited to bone marrow suppression.
* History of malignant tumors, except for basal cell carcinoma, papillary thyroid carcinoma, and various in situ cancers.
* Acute exacerbation of important organ diseases (such as but not limited to chronic obstructive pulmonary disease, coronary heart disease, and renal insufficiency) and/or severe acute infectious diseases (such as but not limited to hepatitis, pneumonia, and myocarditis), American Society of Anesthesiologists score > 3 points.
* Mental disorders, illiteracy, or language communication barriers that prevent the understanding of the study protocol.
* Peripheral sensory neuropathy, unable to receive oxaliplatin-based chemotherapy.
* Continuous use of glucocorticoids for more than 3 days within 1 month prior to signing the informed consent form, or having comorbidities requiring the use of glucocorticoid therapy.
* Unable to undergo enhanced CT examination
* Pregnancy or lactation.
* Refused to participate in this study.
* Other situations in which the researcher deems unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
pCR | 3-5 days of postoperative pathological examination
  the proportion of tumor regression grades 0 (TRG0, disappearance of tumor cells) in the pathological specimens of surgically resected tumors.

SECONDARY OUTCOMES:
R0 resection | 3-5 days of postoperative pathological examination
  the rate of a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.
Disease-free survival (DFS) | From date of the patient signs the informed consent form until the date of earliest occurrence of the patient's tumor recurrence or death, whichever came first, assessed up to 36 months.
  3-year disease-free survival
Overall survival (OS) | From the date of the patient signs the informed consent form until the date of the patient's death, assessed up to 36 months.
  3-year overall survival
Adverse events (AEs) | up to half a year
  the rate of adverse events
Immune-related adverse events (irAEs) | up to half a year
  the rate of immune-related adverse events
Surgical complication | From the day of surgery to 30 days after the operation, including intraoperative and postoperative complications.
  the rate of surgical complication during or after operation.
T lymphocyte | up to 3 months after surgery.
  Cells with cellular immune function. The types and counts of T cells are analyzed using flow cytometry.
Gene mutation signatures of colon cancer | up to 3 months before surgery
  Next-generation target sequencing is performed to analyze the gene mutation signatures.

CONTACTS AND LOCATIONS:
Overall Officials: Sen Zhang, Study Director — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No